CLINICAL TRIAL: NCT05247983
Title: The First Affiliated Hospital of Harbin Medical Uniersity
Brief Title: Tension-free Repair of Inguinal Hernia With "Undissociate Spermatic Cord"
Status: Completed | Type: Observational
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Zhao Lei, Deputy Chief Physician, Harbin Medical University
Other Study IDs: 81902421
Record Dates: First submitted 2022-01-21; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Inguinal Hernia, Without Mention of Obstruction or Gangrene
Keywords: Undissociate Spermatic cord; Inguinal hernia; Hernia exclusion; Hernial sac
MeSH Terms: conditions — Hernia, Inguinal; Gangrene

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: Tension-free repair of inguinal hernia with "Undissociate Spermatic cord"
  Interventions: Procedure: Tension-free repair of inguinal hernia with "Undissociate Spermatic cord"
- control group: Tension-free repair of inguinal hernia with traditional method

INTERVENTIONS:
Procedure: Tension-free repair of inguinal hernia with "Undissociate Spermatic cord" — patient undergoing Tension-free repair of inguinal hernia with "Undissociate Spermatic cord"
  Groups: experimental group

SUMMARY:
The theory of "undissected Spermatic cord (US)" only transected the hernia ring ends in the abdominal cavity, the hernia ring, hernia sac and spermatic cord will not be dissected. Its significance lies in that inguinal hernia repair can get rid of the "entanglement" of hernia sac and spermatic cord and fundamentally change the treatment mode of hernia ring and hernia sac.

DETAILED DESCRIPTION:
In recent years, with the deepening of the anatomical cognition of the inguinal region and the renewal of the hernia repair concept, inguinal hernia repair has become increasingly mature surgical approach. However, no matter how the hernia repair modes change, the treatment and repair of the hernia ring has always been the focus, so that the treatment of the hernia sac has been neglected. From March 2014 to May 2019, there were 132 patients underwent inguinal hernia repair with "Undissociate Spermatic cord" theory (Undissected Spermatic cord and hernia sac, hernia ring and sac exclusion). All the patients were followed up for 18~63 months (mean of 41.5 months) without recurrence. Its significance lies in that inguinal hernia repair can get rid of the "entanglement" of hernia sac and spermatic cord and fundamentally change the treatment mode of hernia ring and hernia sac.

ELIGIBILITY:
Inclusion Criteria:

* Inguinal hernia patients who can tolerate surgery

Exclusion Criteria:

* Patients who cannot tolerate surgery

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inguinal hernia patients
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
surgery time | 0-120minutes
  the operation time
Bleeding | surgery
  Blood loss
hospital stay | 1-30days
  the hospitalization time
Does it recur | 18-63months
  Does it recur

IPD SHARING:
Plan to Share IPD: No